CLINICAL TRIAL: NCT06894693
Title: A Phase I Clinical Trial of RS001 in Patients with Relapsed/Refractory B-Cell Malignancies:
Brief Title: A Phase I Clinical Trial of RS001 in Patients with Relapsed/Refractory B-Cell Malignancies
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Ruishun Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RS001-BCM001
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: B-cell Non-Hodgkin's Lymphoma; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Lymphoma, B-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RS001 injection (Experimental): The trial is divided into two parts: Part A is a dose escalation trial with three dose groups (5×10^6 CAR+ cells/kg, 1×10^7 CAR+ cells/kg and 2×10^7 CAR+ cells/kg at day 0), with 7-18 patients planned to be enrolled. Part B is a dose-expansion trial in which 6~12 patients will receive RS001 infusions at RP2D dose levels.
  Interventions: Biological: RS001 injection

INTERVENTIONS:
Biological: RS001 injection — CD19-CAR-mbIL15-DNT Cells.

SUMMARY:
This study is an open-label, single-arm, dose-escalation and dose-expansion study to evaluate the safety, maximum tolerated dose, pharmacokinetic profile in the body after infusion of RS001 injection, and preliminary efficacy in subjects with CD19-positive relapsed/refractory B-cell malignancies (BCM).

DETAILED DESCRIPTION:
CD19-positive relapsed/refractory B-cell malignancies (including B-cell non-Hodgkin lymphoma, B-cell acute lymphoblastic leukemia).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign an ICF and expect to complete the subsequent follow-up.
2. Aged 18 to 75 years (including cut-offs), regardless of gender.
3. Meet one of the following B-cell malignancies:

<!-- -->

1. . B-cell non-Hodgkin's lymphoma diagnosed as CD19-positive by cytology or histopathology according to WHO 2022 criteria, including pathologically confirmed (1) diffuse large B-cell lymphoma, non-specific type (DLBCL, NOS); (2) follicular lymphoma histopathologically graded as grade 3b (FL3b); (3) follicular lymphoma with diffuse large B-cell transformation; (4) primary mediastinal large B-cell lymphoma (PMBCL); (5) high-grade B-cell lymphoma (HGBCL).

   1. Relapsed/refractory B-cell non-Hodgkin lymphoma, defined as meeting one or more of the following criteria:

      - Definition of relapse: Relapse after achieving remission (PR and CR) with second-line or higher therapy;
      * Definition of refractory: No response to second-line or more therapy: The best efficacy of last therapy is PD or SD (SD requires at least 2 cycles of treatment); Recurrence (must have biopsy-proven recurrence) or progression within 12 months of autologous stem cell transplantation (ASCT) . If salvage therapy, no response to last therapy (SD or PD).
   2. Subjects must have received adequate treatment in the past, which should include the following treatments:

      * Anti-CD20 monoclonal antibody, unless the investigator determines that the tumor is CD20 negative;
      * Chemotherapy containing anthracycline drugs;
      * For subjects with transformed follicular lymphoma (tFL) who have been previously treated with follicular lymphoma (FL) chemotherapy and with transformation to DLBCL show refractory to chemotherapy.
   3. ECOG performance status 0 to 1.
   4. The presence of a measurable lesion that meets one of the following criteria:

      * The long axis of the lymph node lesion exceeds 15 mm in length (the short axis is measurable);
      * The long and short axes of the extralymph node lesion exceed 10 mm in length.
2. Relapsed/refractory B-cell acute lymphoblastic leukemia must meet the following requirements:

   1. Relapsed: Recurrence within 12 months after the first remission;
   2. Refractory: i. failure to remit after more than 6 weeks of induction therapy or failure to remit after two courses of induction therapy; ii. relapse after 2 or more CRs; iii. first relapse after chemotherapy and failure to remit after having received at least 1 salvage therapy; iv. relapse after autologous hematopoietic stem cell transplantation;
   3. Prior to screening, leukemia cells expressing CD19 are detectable in bone marrow or peripheral blood.
   4. Ph+ ALL patients who have failed treatment with at least 2 tyrosine kinase inhibitor (TKI) drugs (including at least 1 2nd generation TKI drug) or are intolerant of drug-related side effects such as allergy to components of the TKI class of drugs, blood abnormalities, liver or kidney impairment, severe cardiovascular toxicity, and other drug-related side effects that prevent them from continuing to be a user; If the patient has the T315I mutation, TKI salvage therapy is not required;
   5. The proportion of primitive and naïve lymphocytes in bone marrow during the screening period ≥5%; 4. Laboratory results within 7 days prior to Lymphodepletion need to meet the following criteria:

   <!-- -->

   1. Coagulation function:

      - Activated partial thromboplastin time ≤ 1.5 times the upper limit of normal (ULN);

      - Prothrombin time (PT) ≤ 1.5 times ULN;
   2. Liver function:

      - Glutathione aminotransferase (AST) ≤ 5 times the upper limit of normal (ULN);

      - Total bilirubin ≤ 1.5 times ULN, unless the subject has documented Gilbert syndrome;

      - Subjects with Gilbert-Meulengracht syndrome with total bilirubin ≤ 3.0 times ULN and direct bilirubin ≤ 1.5 times ULN may be included.
   3. Renal function: Serum creatinine ≤ 1.5 times ULN or a creatinine clearance ≥ 60 ml/min;
   4. Complete blood count (No blood transfusion treatment received within 7 days prior to examination):

      - Haemoglobin ≥ 80 g/L;

      - Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L;
      * A platelet count ≥ 50 x 10^9/L;
   5. Cardiopulmonary function:

      * Left ventricular ejection fraction (LVEF) ≥ 45%;
      * Oxygen saturation ≥ 91%; 5. Female subjects with of childbearing potential should have a negative pregnancy test during the screening period. Any male and female subjects of childbearing potential must agree to use an effective contraception method for at least six months from the time that they sign the informed consent form until the end of the cell infusion. Female subjects without childbearing potential (meeting at least 1 of the following criteria) is described below:

   a. Have undergone a hysterectomy or bilateral oophorectomy; b. Medically recognised ovarian failure; c. Medically recognised as post-menopausal (at least 12 consecutive months of menopause without pathological or physiological cause).

Exclusion Criteria:

1. Other malignancies within 5 years prior to screening, except adequately treated carcinoma in situ of the cervix, basal cell or squamous epithelial cell skin cancer, post-radical localized prostate cancer, post-radical ductal carcinoma in situ, and post-radical thyroid cancer;
2. Any unstable systemic disease: including but not limited to active infection (other than local infection), unstable angina, cerebrovascular accident or transient ischaemia (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), New York Heart Association class III or IV cardiac insufficiency, refractory hypertension (refractory hypertension is defined as blood pressure that has not reached standard after >1 month of reasonably tolerable treatment with ≥3 antihypertensive drugs (including diuretics) at adequate doses based on lifestyle improvement or blood pressure that is not effectively controlled with ≥4 antihypertensive drugs), severe cardiac arrhythmias requiring pharmacologic treatment, hepatic arrhythmias, liver diseases, kidney diseases or metabolic disorders;
3. Patients with B-cell non-Hodgkin's lymphoma with active central nervous system invasion.
4. Patients with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and peripheral blood hepatitis B virus (HBV) DNA titres not within the normal reference range, positive hepatitis C virus (HCV) antibody and peripheral blood HCV RNA ,positive for human immunodeficiency virus (HIV), or positive for cytomegalovirus (CMV) DNA, or positive syphilis test.
5. Subjects who are receiving systemic steroids prior to screening and who are judged by the investigator to require long-term treatment with systemic steroids during the treatment period (except for inhaled or topical use).
6. Previous organ transplantation or preparation for organ transplantation (except for haematopoietic stem cell transplantation).
7. Persons with acute/chronic Graft-vs-Host Disease (GvHD).
8. Patients have received a haematopoietic stem cell transplant within 2 months prior to screening.
9. Patients who have previously received any CD19-CAR-T/NK cell therapy, or received CAR-T/NK cell therapy targeting other antigens within the three months prior to screening.
10. Active neurological autoimmune or inflammatory diseases (e.g. Guillain-Barre Syndrome (GBS), Amyotrophic lateral sclerosis (ALS)).
11. Clinically significant active cerebrovascular diseases (such as cerebral edema, posterior reversible encephalopathy syndrome).
12. Patients with a life expectancy of less than 3 months.
13. Participants who have previously been involved in other interventional clinical studies and received active investigational drugs, with the last use of an unapproved new drug being less than 28 days prior to signing the informed consent for this trial, or the last use of an approved drug being less than five half-lives prior to cell infusion.
14. Received attenuated live vaccine within 6 weeks prior to lymphodepletion.
15. The subjects have contraindications or hypersensitivity reactions to fludarabine, cyclophosphamide, tocilizumab, investigational product and its ingredients.
16. Remaining within the washout period of other antitumor treatments prior to lymphodepletion.
17. Patients who, in the investigator's judgment and/or clinical criteria, have a contraindication to any of the study procedures or have other medical conditions that may place them at unacceptable risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | Up to 28 days
  To evaluate the safety, tolerability, and determine the recommended dosage of RS001 for BCM subjects.
Maximum Tolerated Dose (MTD) | Up to 28 days
  MTD is the highest dose for DLT in ≤1/6 subjects.
Incidence of abnormalities | Up to 28 days
  Incidence of abnormalities in AE/SAE/AESI/laboratory tests/electrocardiograms/vital signs.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) indicator (Cmax) | Up to 90 days
  The peak concentration of CD19-CAR-mbIL15-DNT cells amplified in the peripheral blood (Cmax, detected by qPCR or Flow Cytometry).
Pharmacokinetics (PK) indicator (AUC) | Up to 90 days
  CD19-CAR-mbIL15-DNT cells blood concentrations will be measured at different time points to evaluate the area under the curve (AUC). (AUC, detected by qPCR or Flow Cytometry).
Pharmacokinetics (PK) indicator (Tmax) | Up to 90 days
  CD19-CAR-mbIL15-DNT cells blood concentrations will be measured at different time points to evaluate the peak plasma time (Tmax). Tmax is defined as the time to reach the highest concentration (Tmax, detected by qPCR or Flow Cytometry).
Pharmacokinetics (PK) indicator (T1/2) | Up to 90 days
  CD19-CAR-mbIL15-DNT cells blood concentrations will be measured at different time points to evaluate the elimination half-life in hours (T1/2). T1/2 is defined as the time point when the concentration of CD19-CAR-mbIL15-DNT reaches half of maximum in a patient's peripheral blood (T1/2, detected by qPCR or Flow Cytometry).
Overall Response Rate | Up to 2 years
  Objective response rates (ORR; complete response [CR] + partial response [PR]) in B-NHL subjects and composite complete remission rates (CRc; CR + CR with incomplete hematologic recovery [CRi]) in ALL subjects were assessed using Lugano 2014 criteria / LYRIC Criteria (2016) and National Comprehensive Cancer Network (NCCN) guidelines (v3.2025), respectively.
Disease Control Rate | Up to 2 years
  The percentage of PR, CR and SD patients in the total B-NHL patient population.
Duration of Response | Up to 2 years
  The time from the start of the first assessment of CR or PR to the first assessment as disease recurrence or progression or death in B-NHL subjects.
  The time from the first assessment of the tumor for CR or CRi to the first assessment of disease recurrence or death from any cause in B-ALL subjects.
Progression Free Survival | Up to 2 years
  The time from the first cell infusion to the first evaluation of tumor progression or death from any cause in B-NHL subjects.
Overall Survival | Up to 2 years
  From the date of entry into the clinical study until death from any cause
Overall Response Rate at 3 months | Up to 3 months
  The percentage of PR and CR patients in B-NHL patient population at 3 months.
Relapse-Free Survival | Up to 2 years
  Evaluate only ALL patients who achieved CR or CRi. This refers to the period from the first assessment of CR or CRi until the first evaluation indicating disease relapse or death from any cause during CR or CRi.
Event-Free Survival | Up to 2 years
  This is used for evaluating all ALL subjects. The period starts from the first infusion of RS001 injection until treatment failure, relapse, or death (any cause), whichever occurs first. For subjects without these events, the timeframe will be calculated up to the date of the last follow-up visit. For patients who did not achieve CR or CRi, EFS will be calculated from the clinical trial enrollment date until disease progression or death, with the first occurring event being considered as the endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: JunYuan Qi, MD, PHD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China